CLINICAL TRIAL: NCT05875532
Title: Incidence Probability of Progression to Progressive Fibrosing Interstitial Lung Diseases and Status of Management and Treatments in Patients With Fibrosing Interstitial Lung Diseases Other Than Idiopathic Pulmonary Fibrosis in Japan
Brief Title: Study of Progression to Progressive Fibrosing Interstitial Lung Disease (PF-ILD) Incidence/Management and Treatment
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0523
Record Dates: First submitted 2023-04-30; First posted 2023-05-25 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with an ILD other than IPF: Patients in Japan with data available in the Medical Data Vision (MDV) database, presenting an underlying pre-specified Interstitial Lung Disease (ILD) between 01-Jan-2012 to 28-May-2020 and received a second diagnosis of a fibrosing ILD other than Idiopathic Pulmonary Fibrosis (IPF) in the period of 01-Jan-2013 to 6 months before 28-May-2020.

SUMMARY:
The primary objective for this trial is to investigate the incidence probability of progression to Progressive Fibrosing Interstitial Lung Diseases (PF-ILDs) in patients with fibrosing ILD other than Idiopathic Pulmonary Fibrosis (IPF) in real-world setting in Japan.

The secondary objective is to investigate the characteristics of procedures for management and treatment in patients with fibrosing ILD other than IPF in real-world setting in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with at least two fibrosing Interstitial Lung Disease (ILD) codes on different dates in the patient identification period
2. Patients aged 18 years and older on the index date
3. Patients for whom data for the 12 months prior to the index date can be extracted as baseline data

Exclusion Criteria:

1. Patients grouped into the underlying disease of Idiopathic Pulmonary Fibrosis (IPF)
2. Patients who have met PF-ILD progression criteria during the baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with at least two fibrosing ILD codes (International Statistical Classification of Diseases and Related Health Problems (ICD-10) code or disease code)
Sampling Method: Non-Probability Sample
Enrollment: 34960 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boehringer Ingelheim Pharmaceuticals, Inc., Ridgefield, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective cohort study using the Medical Data Vision (MDV) database to study progression to Progressive Fibrosing Interstitial Lung Disease (PF-ILDs) in a real-world setting in Japan. Data was extracted for the period of 01-Jan-2012 to 28-May-2020 for patients presenting pre-specified ILDs that received a second diagnosis of a fibrosing ILD other than Idiopathic Pulmonary Fibrosis (IPF) between 01-Jan-2013 to 6 months before 28-May-2020.
Pre-assignment Details: Patients that met all inclusion criteria and none of the exclusion criteria were followed from the day after of the second diagnosis of a fibrosing ILD other than IPF - index date - until the end of study period (28-May-2020), the last encounter in the MDV database or in-hospital death, whichever occurs first.
Period: Overall Study
Arm/Group | Patients With an ILD Other Than IPF
Started | 34960
Completed | 34960
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set: Patients in Japan with data available in the Medical Data Vision (MDV) database, between 01-Jan-2012 to 28-May-2020, who met all inclusion criteria and none of the exclusion criteria.
Arm/Group | Patients With an ILD Other Than IPF
Number analyzed (Participants) | 34960
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at the second diagnosis of a fibrosing ILD other than IPF - index date
  Years | 71.13 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16597
  Male | 18363
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Probability of Progression to Pulmonary Fibrosing-Interstitial Lung Disease (PF-ILDs)
Description: The cumulative incidence probability is the estimate of the risk a patient will experience by 6, 12, 18 and 24 months after the second diagnosis of fibrosing ILD (index date) of progression to PF-ILDs. It is the complement of the Kaplan-Meier estimates. The Greenwood's variance estimate was used to calculate the 95% confidence interval.
  Disease progression was defined as 3 or more pulmonary function tests within 365 days, 3 or more tomographies within 365 days, 1 or more claims for oxygen therapy during follow-up, 1 or more respiratory hospitalizations during follow-up, 1 or more claims for palliative care during follow-up, 1 or more lung transplant during follow-up, 1 or more claims for immunosuppressive drugs during follow-up, 1 or more claims for oral corticosteroid during follow-up, and 1 or more claims for Nintedanib during follow-up. Follow-up was between 1-Jan-2013 to 28-May-2020, the last encounter in Medical Data Vision database, or in-hospital death, whichever occurs first.
Time Frame: At 6, 12, 18 and 24 months after the index date, defined between 01-Jan-2013 and 6 months before 28-May-2020
Population: Full analysis set: Patients in Japan with data available in the Medical Data Vision (MDV) database, between 01-Jan-2012 to 28-May-2020, who met all inclusion criteria and none of the exclusion criteria. The number of patients analyzed displays the number of patients at risk of progression at the time of interest.
Measure: Number (95% Confidence Interval); unit: Cumulative incidence probability
Arm/Group | Patients With an ILD Other Than IPF
Number analyzed (Participants) | 34960
Cumulative incidence probability
  6 months: number analyzed (Participants) | 27770
  6 months | 0.147 [0.143 to 0.151]
  12 months: number analyzed (Participants) | 20888
  12 months | 0.249 [0.244 to 0.253]
  18 months: number analyzed (Participants) | 15921
  18 months | 0.334 [0.329 to 0.34]
  24 months: number analyzed (Participants) | 12117
  24 months | 0.395 [0.389 to 0.401]

2. Secondary Outcome: Number of Patients With Treatment of Interest During Follow-up Period
Description: Number of patients treated with immunosuppressive drugs (Rituximab, Tacrolimus, Mycophenolate, Cyclosporine, Cyclophosphamide, Azathioprine, Tocilizumab), oral corticosteroids, or nintedanib during the follow-up period. The follow-up period was between the second diagnosis of a fibrosing ILD (index date) and end of study (28-May-2020), the last encounter in Medical Data Vision database, or in-hospital death, whichever occurs first.
Time Frame: Up to 7.43 years, from 01-Jan-2013 to 28-May-2020
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With an ILD Other Than IPF
Number analyzed (Participants) | 34960
Participants
  Rituximab | 49
  Tacrolimus | 499
  Mycophenolate | 30
  Cyclosporine | 200
  Cyclophosphamide | 225
  Azathioprine | 201
  Oral corticosteroid | 2065
  Tocilizumab | 46
  Nintedanib | 472

3. Secondary Outcome: Number of Patients With Management of Interest During Follow-up Period
Description: Number of patients with oxygen therapy (HOT), lung transplant and palliative care (oxygen inhalation, opioid use) as disease management during the follow-up period. The follow-up period was between the second diagnosis of a fibrosing ILD (index date) and end of study (28-May-2020), the last encounter in Medical Data Vision database, or in-hospital death, whichever occurs first.
Time Frame: Up to 7.43 years, from 01-Jan-2013 to 28-May-2020
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With an ILD Other Than IPF
Number analyzed (Participants) | 34960
Participants
  Oxygen therapy (HOT) | 1641
  Lung transplant | 0
  Palliative care (oxygen inhalation, opioid use) | 9520

ADVERSE EVENTS:
Time Frame: Adverse event information was not applicable for this study.
Description: As this is a non-interventional study with secondary use of data retrieved from Medical Data Vision database, safety monitoring and safety reporting on an individual case level is not applicable. All-Cause Mortality, Serious Adverse Events and Other Adverse Events are not collected in the database. "0" total Number of Participants at Risk means "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Arm/Group | Patients With an ILD Other Than IPF
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The Medical Data Vision (MDV) database did not have pulmonary function test results and there was no evidence of using claims data to define the events fibrosing Interstitial Lung Disease (ILD) patients other than Idiopathic Pulmonary Fibrosis (IPF) and progression to Progressive Fibrosing Interstitial Lung Diseases (PF-ILDs) in the validated algorithm. Data generated in the clinics/hospitals other than hospitals included in the MDV database were not captured.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT05875532/Prot_SAP_000.pdf